CLINICAL TRIAL: NCT05765526
Title: A Novel Electrolyzed Water Spray Reduces Discomfort or Itching Scores of Patients With Scalp Discomfort or Itching: A Clinical Study
Brief Title: A Novel Electrolyzed Water Spray Treatment for the Discomfort or Itching of Patients With Scalp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jia19961125
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-02

CONDITIONS: Scalp Dermatoses
Keywords: Electrolyzed water device; Hydroxyl radical; Tap water; Spray; Scalp discomfort; Scalp itching
MeSH Terms: conditions — Scalp Dermatoses

STUDY DESIGN:
Intervention Model Description: An open label, single arm and before and after treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The scalp of discomfort or itching and one treatment (Experimental): Participants with discomfort or itching scalp who will receive one treatment with the device and complete the questionnaire.
  Interventions: Device: A novel electrolyzed water spray

INTERVENTIONS:
Device: A novel electrolyzed water spray — Study staff will use the novel electrolyzed water spray device and spray for approximately 10 minutes on the participant's scalp until half bottle (200ml) of water is used. Their scalp will then be rinsed and gently dried with a towel.

SUMMARY:
The purpose of this study is to test whether the reduction of the discomfort or itching with the scalp of patients by use of the novel electrolyzed water spray will produce improvement in the condition of the scalp.

DETAILED DESCRIPTION:
In this study, water inculding tap water,pure water and salt water, and an apparatus for producing electrolyzed water (https://www.deposon.com.cn; https://www.deposon.com）were used to generate an electrolyzed water mist spray or spray. This instantly generated electrolyzed water mist spray or spray has oxidation-reduction potential (ORP) ≥1200mv,and contains non-specific total oxidation capacity which equals to 0.28±0.10ppm,0.06±0.04ppm and 3.92±0.39ppm of desolved ozone. This instantly generated electrolyzed water mist spray or spray does not release detectable ≥0.1mg/m3 of gaseous ozone. This instantly generated electrolyzed water mist spray or spray has pH 8.4±0.4 and releases negative air ion.The apparatus for producing electrolyzed water has a positive electrode which is covered by a conductive diamond material (Patent# CN215308550U). This is an open-label, single-arm and before and after treatment comparison study. In this study, this novel electrolyzed water device and the water spray are used to treat scalp itching. The reduction in the scalp of discomfort or itching evaluation and adverse event assessments will be performed at each visit. Safety analysis will be assessed based on the reports of adverse events during the study.

ELIGIBILITY:
Inclusion Criteria:

* The patients with scalp discomfort or itching

Exclusion Criteria:

* severe scalp discomfort or itching; 80 years or elder

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
A discomfort or itching scale made by modifing a pain scale (NPRS) | 5 days
  This Score is based on descriptions of the discomfort or itching that patients rate 0-10 to assess the condition of their scalp. A higher score means a worse outcome. 0 means "no discomfort or itching " and 10 means "the most discomfort or itching".

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: until publication of this clinical study and international patent granted